CLINICAL TRIAL: NCT00005091
Title: A Phase II Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Patients With Stage IIIb or Stage IV Non-Small Cell Lung Cancer as First Line Therapy
Brief Title: DX-8951f in Treating Previously Untreated Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: DAIICHI-8951E-PRT017; CDR0000067724 (Registry Identifier: PDQ (Physician Data Query)); EU-99044
Record Dates: First submitted 2000-04-06; First posted 2004-06-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-01

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DX-8951f in treating patients who have previously untreated stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of DX-8951f in previously untreated patients with stage IIIB or IV non-small cell lung cancer. II. Evaluate the quantitative and qualitative toxic effects of this regimen in these patients. III. Evaluate the pharmacokinetics of this regimen in these patients. IV. Assess the time to progression and survival status of these patients.

OUTLINE: This is a multicenter study. Patients receive DX-8951f IV over 30 minutes daily for 5 days. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for survival.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed unresectable, metastatic, or recurrent non-small cell lung cancer Stage IIIB or IV Measurable disease No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT or SGPT no greater than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present) Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No active congestive heart failure Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No concurrent serious infection No other malignancy within past 5 years except nonmelanomatous skin cancer No overt psychosis, mental disability, or incompetence No life threatening illness

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to greater than 25% of the bone marrow No concurrent radiotherapy Surgery: No concurrent surgery Other: At least 28 days since prior investigational drugs No other concurrent investigational drugs during or within 28 days after final dose of study drug No concurrent drugs that induce or inhibit CYP3A enzyme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Thatcher, PhD, FRCP, Study Chair — The Christie NHS Foundation Trust
Locations (6):
- Helsinki University Central Hospital, Helsinki, Finland
- Thoraxklinik Rohrbach, Heidelberg, Germany
- Ospedale Bellaria, Bologna, Italy
- Academisch Ziekenhuis der Vrije Universiteit, Amsterdam, Netherlands
- United Kingdom (2):
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Oxford Radcliffe Hospital, Oxford, England

REFERENCES:
- [Result] Braybrooke JP, Ranson M, Manegold C, Mattson K, Thatcher N, Cheverton P, Sekiguchi M, Suzuki M, Oyama R, Talbot DC. Phase II study of exatecan mesylate (DX-8951f) as first line therapy for advanced non-small cell lung cancer. Lung Cancer. 2003 Aug;41(2):215-9. doi: 10.1016/s0169-5002(03)00190-9. PMID 12871785